CLINICAL TRIAL: NCT06440746
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled, Multicenter Phase 2/3 Study of Efficacy and Safety of Olokizumab in Subjects With Progressive Fibrosing Interstitial Lung Diseases
Brief Title: Efficacy and Safety of Olokizumab in Patients With Progressive Fibrosing Interstitial Lung Diseases
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: R-Pharm International, LLC (Industry)
Collaborators: R-Pharm (Industry); Exacte Labs LLC (Industry); Data Management 365 (Industry); Keystat, LLC (Industry)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL04041109
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Lung Diseases, Interstitial
Keywords: Progressive Fibrosing Interstitial Lung Diseases; Olokizumab; Forced vital capacity
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1:OKZ 64 mg q4w (Experimental): SC injections of OKZ 64 mg q4w
  Interventions: Drug: Subcutaneous (SC) injections of OKZ 64 milligrams (mg) every 4 weeks (q4w), one injection of 0.4 millilitre (mL)
- Arm2:Placebo (Placebo Comparator): SC injections of Placebo q4w
  Interventions: Drug: SC injections of Placebo every 4 weeks (q4w), one injection of 0.4 mL

INTERVENTIONS:
Drug: Subcutaneous (SC) injections of OKZ 64 milligrams (mg) every 4 weeks (q4w), one injection of 0.4 millilitre (mL) — Olokizumab is a sterile solution for subcutaneous injection in a 2-mL clear Type I glass vial, containing a target fill volume of 0.5 mL (for withdrawal of no less than 0.4 mL) of olokizumab drug substance at a concentration of 160 milligrams (mg)/mL.
  Other Names: Artlegia
  Arms: Arm1:OKZ 64 mg q4w
Drug: SC injections of Placebo every 4 weeks (q4w), one injection of 0.4 mL — Placebo (sodium chloride 0.9 %) does not contain any active pharmaceutical ingredients. Placebo will be supplied in 2-mL, 5-mL, or 10-mL ampoules made of low-density polyethylene or polypropylene.
  Arms: Arm2:Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of olokizumab (OKZ) compared to placebo in patients progressive fibrosing Interstitial lung diseases (ILD).

DETAILED DESCRIPTION:
This is a phase 2/3 study with double-blind parallel-group adaptive design.

The study will include the following periods:

1. Screening period (4 weeks) Screening period (before the first administration of the test drug). Before being included in the study, patients will be provided with complete information about this clinical trial and signs the Informed consent Form (IF). After that the researcher will decide whether or not the patient can be randomized into the study.
2. Double-blind Treatment period (48 weeks). Following the completion of a Treatment period, all patients will be enrolled in Follow-up Period (FU).
3. Follow-up Period (24 weeks). During the FU Period, patients will visit study sites after 4,12 and 24 weeks after the end of the Treatment Period to complete FU-1 (Week 52), FU-2 (Week 60) and FU-3 (Week 72) visits.

The overall study duration for the patients will be approximately 76 weeks (including the 4 weeks screening period)

The analysis will be conducted in two sequential steps:

* the interim analysis after 61 percent (%) of patients have completed the Treatment period (not including the FU period)
* the final analysis when all patients have completed all periods (the Treatment and the FU periods).

ELIGIBILITY:
Inclusion Criteria:

1. The patient has signed the Informed Consent Form
2. Progressive fibrosing ILD confirmed by high-resolution computed tomography (HRCT) documented evidence of >10% lung tissue affected at Screening:

   A. Patients with an usual interstitial pneumonia (UIP) -like radiological pattern described in the 2022 American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American Thoracic Association guidelines for the management Idiopathic pulmonary fibrosis (IPF) that do not have an identified primary condition

   В. Patients with progressive interstitial pneumonia with autoimmune features (IPAF) as defined in the American Thoracic Society/European Respiratory Society Statement, 2015

   С. Patients with progressive lung fibrosis associated with different disorders (c) such as systemic connective tissue diseases, chronic fibrosin hypersensitivity pneumonitis (HP), idiopathic non-specific interstitial pneumonia (iNSIP) or sarcoidosis.

   Disease progression will be established based on a combination of criterion (I)(a) and criterion (II) or criterion (III)(b)

   I. Clinically significant decrease in FVC% predicted defined as absolute decrease of ≥ 5% within 12 months prior to screening or an absolute decrease DLCO (corrected for hemoglobin) of ≥10% predicted within 12 months prior to screening.

   II. Worsening respiratory symptoms without an alternative explanation within 12 months prior to screening.

   III. Increased area affected with fibrosis on chest HRCT (b) (according to the 2022 American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American Thoracic Association guidelines) within 24 months prior to screening.
   1. To assess this criterion (I), patient's pulmonary function test (PFT) results obtained within 12 months prior to screening must available. If data from multiple PFTs are available, the earliest results must be used for assessment.
   2. Patients' results of at least one chest HRCT investigation performed no earlier than 24 months before randomization must be available for review. If results of multiple HRCT examinations are available, patient eligibility must be based on the earliest results.
   3. stable course of the main disease not requiring a change in maintenance treatment.
3. ILD duration of no more than 8 years from the onset of respiratory symptoms by the date screening begins.
4. Elevated acute phase reactants at screening not related to other causes:

   C-reactive protein level ≥6 mg/l or Erythrocyte Sedimentation Rate (ESR) ≥28 millimeters per hour (mm/hour).
5. FVC ≥ 45% and ≤ 80% predicted at screening.

Non-Inclusion Criteria:

1. Hemoglobin-corrected DLCO < 30% predicted at screening.
2. Significant airway obstruction at screening defined as a Forced expiratory volume in 1 second (FEV1) / FVC ratio of <70 %.
3. Use of interleukin-6(IL-6 )inhibitors or IL-6 receptor inhibitors except for CoronaVirus Disease2019 (COVID-19) treatment. If those medications are used to treat COVID-19, the last administration of IL-6 inhibitors or IL-6 receptor inhibitors must have occurred at least 6 months prior to screening.
4. Administration of rituximab within less than 12 months prior to screening.
5. Treatment with systemic glucocorticosteroids (GCS) at >10 mg/day calculated for prednisolone; or a change in the dose of GCS within 4 weeks before/during the screening period; or planned dose changes during the trial.
6. A history of bone marrow transplantation, total lymphoid tissue irradiation, or administration of ablative ultra-high doses of cyclophosphamide.
7. Initiation of mycophenolate mofetil or antifibrotic agents (for patients receiving mycophenolate mofetil and/or antifibrotics at study entry) less than 12 months prior to screening.

   • If a patient has been taking antifibrotic drugs for <12 months and ≥6 months, and the spirometry/Diffusion Capacity Of The Lungs For Carbon Monoxide (DLCO) used to assess progression was performed within ±2 weeks of actually starting antifibrotic drugs, the patient may be included in the study
8. Discontinuation of previously prescribed antifibrotic agents within 6 months prior to screening (for patients not receiving antifibrotic drugs at study entry).
9. Participation in any other clinical trial less than 30 days prior to the baseline assessment or less than 5 half-lives of the medication examined in another clinical trial, whichever is longer.
10. Laboratory abnormalities as follows:

    * Alanine Aminotransferase (ALT) or Aspartate Aminotransferase(AST) ≥ 1.5×Upper Limit Normal (ULN)
    * Platelet count <100×10^9/litre (l) (<100000/cubic millimetre (mm^3)
    * Leukocyte count <3.5×10^9/l
    * Absolute neutrophil count <2000×10^6/l (<2000/mm^3).
11. Concurrent malignancy or a history of malignancy within the last 5 years.
12. Any acute infection at screening or exacerbation of a chronic infection, any infection requiring oral antibiotics or antivirals within 4 weeks prior to screening, injection of antimicrobial agents within 6 weeks before randomization, severe or recurrent infections requiring hospital admission within 6 months before randomization.
13. Patients with evidence of disseminated herpes zoster infection, herpes zoster with encephalitis, meningitis, or other forms of herpes zoster infection that do not resolve without treatment and occurred within 6 months prior to screening.
14. Evidence of any other chronic infection (including sepsis, invasive fungal infection, histoplasmosis, osteomyelitis) which, in the opinion of the Investigator, may increase the risk of infectious complications during the trial.
15. Patients with diverticulitis or other symptomatic gastrointestinal diseases that may lead to perforation, including such history (for example, diverticulitis, gastrointestinal perforation, ulcerative colitis).
16. Women of child-bearing potential or men whose partners are women of child-bearing potential who do not want to use highly effective methods of contraception during the trial and for at least 3 months after the last administration of the investigational product.
17. Known hypersensitivity to OKZ or any other component of the product or placebo.
18. History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies.
19. Other protocol-defined non-inclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2027-04-09 (Estimated); Study Completion 2028-12-25 (Estimated)

PRIMARY OUTCOMES:
The rate of forced vital capacity (FVC) | 48 weeks
  FVC decline rate assessed over 48 weeks of therapy. FVC is the maximum amount of air that can be exhaled when blowing out as fast as possible.

SECONDARY OUTCOMES:
Change in FVC from baseline | 24, 48 weeks.
  Absolute change in FVC from baseline at treatment weeks 24 and 48.
Change in FVC.% predicted | 24,48 weeks
  Change in FVC% predicted from baseline at treatment weeks 24 and 48.
Number of patients (in %) with a decrease in FVC | 48 weeks
  Number of patients (in %) with a decrease in FVC of ≥10 % predicted.at treatment week 48.
Number of patients (in %) with improved pulmonary function | 48 weeks
  Number of patients (in %) with improved pulmonary function (change from baseline in FVC >0% predicted.
Change of Diffusing capacity of the lungs for carbon monoxide (DLCO) | 24,48 weeks
  Change in absolute values of DLCO from baseline at treatment weeks 24 and 48.
Change in the values of quantitative assessment of lung fibrosis from baseline | 48 weeks
  Change in the values of quantitative assessment of lung fibrosis from baseline based on high-resolution computed tomography (HRCT) data at treatment week 48.
Proportion of patients with progression or death | 48 weeks
  Proportion of patients with progression or death: the first event defined as death.
  Progression is a decrease in FVC ≥10% predicted, or decrease in DLCO ≥15% predicted from their baseline values.
Time to progression or death assessed over 48 weeks of treatment | 48 weeks
  Time to progression or death assessed over 48 weeks of treatment.
Time to exacerbation over 48 weeks of treatment | 48 weeks
  An exacerbation of idiopathic lung fibrosis and other ILDs is defined as worsening shortness of breath over the past 30 days combined with evidence of new bilateral lesions appearing as ground-glass opacities and/or consolidations on a chest HRCT scan without other alternative causes (infections and other).
Proportion of patients with exacerbation at treatment weeks 24 and 48 | 24,48 weeks
  Proportion of patients with exacerbation over 48 weeks of treatment.
Change in Functional Assessment of Chronic Illness Therapy (FACIT)-Dyspnea scores from baseline at treatment weeks 24 and 48 | 24,48 weeks
  FACIT-Dyspnea questionnaire includes Dyspnea subscale, that measures the severity of dyspnea when doing everyday activities, and Functional Limitations subscale that measures the amount of difficulty experienced while doing these activities due to dyspnea in the past 7 days. Both subscales contain 10 items scored from 0 (best) to 4 (worst).
  A raw score (normal-worst range 0-30) is calculated as: Sum individual item scores * 10 / number of items answered. Raw scores are then converted to scale scores using the table included in the FACIT Dyspnoea Scale Short Form Scoring Guideline.
  Scale score range: Dyspnea subscale from 27.7 (normal condition) to 75.9 (severe symptoms); Functional Limitations subscale from 29.7 (not limited) to 76.7 (severely limited)
Change in Short Form-36 (SF-36) scores from baseline at treatment weeks 24 and 48 | 24,48 weeks
  36-Item Short-Form Health Survey (SF-36) is a patient reported survey of health consisting of 36 items that taps eight health concepts (domains): vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; mental health. It also includes a single item that provides an indication of perceived change in health. For each domain a scaled score is calculated as the weighted sum of the questions in this section. Each scale is directly transformed into a 0 to 100 scale on the assumption that each question carries equal weight. A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in Modified Medical Research Council ( mMRC) dyspnea score from baseline at treatment weeks 24 and 48 | 24,48 weeks
  Modified Medical Research Council (mMRC) Dyspnea Scale is used to assess perceived degree of baseline functional disability due to dyspnea. Participants indicate a score on 5-point scale according to the severity of their symptoms: none = 0; mild = 1; moderate = 2; severe =3; very severe = 4

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (33):
- Russia (33):
  - Regional Clinical Hospital Regional state budgetary healthcare institution, Barnaul
  - Regional Clinic Hospital№3, Chelyabinsk
  - Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - State budgetary healthcare institution of the Leningrad region "Gatchina Clinical Interdistrict Hospital", Gatchina
  - LLC" Medsi-Izhevsk", Izhevsk
  - LLC "Scientific Research Medical Complex "Your Health", Kazan'
  - Kuzbass Clinical Hospital Emergency Medical Care named after Podgorbunsky M.A, Kemerovo
  - State Budgetary Healthcare Institution Research Institute-Karpaty Clinical Hospital No. 1 named after prof. S.V. Ochapovsky, Krasnodar
  - City Clinical Hospital named after Davydovsky I.V., Moscow
  - GBUZ Moscow Clinical Scientific Center named after Loginov MHD, Moscow
  - Scientific Research Institute of Reumatology named after Nasonova V.A, Moscow
  - Moscow City Polyclinic №52, Moscow
  - Clinical Hospital №4 of Sechenov University, Moscow
  - Clinical Hospital №3 of Sechenov University, Moscow
  - State Budgetary Healthcare Institution of Moscow City "City Clinical Hospital №52" of the Moscow City Health Department", Consultative and diagnostic department №2, Moscow
  - State Budgetary Healthcare Institution of Moscow City "City Clinical Hospital №52" of the Moscow City Health Department", Moscow
  - FSBEI HE "Russian University of Medicine", MoH of Russia, Moscow
  - Moscow Regional Research and Clinical Institute "MONIKI", Moscow
  - Federal Research Center Institute of Cytologyand Genetics,Siberian Branch of Russian Academy of Sciences, Novosibirsk
  - Republican Hospital named after V.A. Baranov, Petrozavodsk
  - Saint-Petersburg State Research Institute of Phthisiopulmonology of the Ministry of Healthcare of the Russian Federation, Saint Petersburg
  - LLC"Energy of Health", Saint Petersburg
  - Medical Center "Interleukin", Saint Petersburg
  - City Multidisciplinary Hospital №2-Expert Center in the field of Pulmonology, Saint Petersburg
  - LLC"Kurator", Saint Petersburg
  - State Healthcare Institution "Regional Clinical Hospital", Saratov
  - Regional state budgetary healthcare institution "Clinical Hospital No. 1", Smolensk
  - Regional State Budgetary Healthcare Institution "Medical and Sanitary Unit No. 2, Tomsk
  - Federal State Budgetary Educational Institution of Higher Education "Bashkir State Medical University" of the Ministry of Health of the Russian Federation, Ufa
  - State Budgetary Healthcare Institution of the Vladimir Region "Regional Clinical Hospital", Vladimir
  - Budgetary healthcare institution of the Voronezh region "Voronezh Regional Clinical Hospital No1", Voronezh
  - Clinical Hospital of Emergency Medical Care named after Solovyov N.V, Yaroslavl
  - Ural research Institute of Phthisiopulmonology, Yekaterinburg